CLINICAL TRIAL: NCT01302899
Title: A Single-blind, Double Dummy, Randomized, Multi-dose, Two Sequence, Crossover, Study to Investigate the Effects of Renin Inhibitor (Aliskiren 300 mg) on Albuminuria in Non-diabetic Nephropathy Patients Treated With Ramipril 10 mg and Volume Intervention (ARIA)
Brief Title: To Study the Effects of Aliskiren on Albuminuria and Various Biomarkers in Patients With Nephropathy
Acronym: ARIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In consequence of termination of ALTITUDE. A number of studies were continued in consultation with the Altitude Data Monitoring Committee.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CSPP100A2260; 2009-012196-10 (EudraCT Number)
Record Dates: First submitted 2011-02-09; First posted 2011-02-24 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Non-diabetic Nephropathy
MeSH Terms: interventions — aliskiren; Hydrochlorothiazide; Ramipril

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)+HCTZ/Ram+Ali/Ram (Experimental): Period 1(Day 1 to end of week 6): 1 tablet ramipril 10 mg once daily (o.d.) + 2 tablets placebo to aliskiren 150mg o.d. + 1 capsule Hydrochlorothiazide (HCTZ) 25 mg o.d.
  Period 2 (Weeks 7 to 12): 1 tablet ramipril 10 mg o.d.+ 1 tablet aliskiren 150 mg in 1st week of period; thereafter, 2 tablets aliskiren 150mg o.d.+ 1 capsule HCTZ 25 mg o.d.
  Period 3 (Weeks 13 to 18): 1 tablet ramipril 10 mg o.d. + 2 tablets aliskiren 150mg o.d. + 1 capsule placebo to HCTZ 25 mg o.d.
  Period 4 (Weeks 19 to 26): 1 tablet ramipril 10 mg o.d. + 2 tablets placebo to aliskiren 150mg o.d. + 1 capsule placebo to HCTZ 25 mg o.d.
  Interventions: Drug: Aliskiren; Drug: Placebo to Aliskiren; Drug: Hydrochlorothiazide (HCTZ); Drug: Placebo to Hydrochlorothiazide (HCTZ); Drug: Ramipril
- Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)/Ram+Ali + HCTZ/Ram (Experimental): Period 1(Day 1 to end of week 6): 1 tablet ramipril 10 mg once daily (o.d.) + 2 tablets placebo to aliskiren 150mg o.d. + 1 capsule Hydrochlorothiazide (HCTZ) 25 mg o.d.
  Period 2 (Weeks 7 to 12): 1 tablet ramipril 10 mg o.d.+ 1 tablet aliskiren 150 mg in 1st week of period; thereafter, 2 tablets aliskiren 150mg o.d.+ 1 capsule placebo to HCTZ 25 mg o.d.
  Period 3 (Weeks 13 to 18): 1 tablet ramipril 10 mg o.d. + 2 tablets aliskiren 150mg o.d. + 1 capsule HCTZ 25 mg o.d.
  Period 4 (Weeks 19 to 26): 1 tablet ramipril 10 mg o.d. + 2 tablets placebo to aliskiren 150mg o.d. + 1 capsule placebo to HCTZ 25 mg o.d.
  Interventions: Drug: Aliskiren; Drug: Placebo to Aliskiren; Drug: Hydrochlorothiazide (HCTZ); Drug: Placebo to Hydrochlorothiazide (HCTZ); Drug: Ramipril

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg (Tablet)
Drug: Placebo to Aliskiren — Aliskiren 150 mg Matching Placebo (Tablet)
Drug: Hydrochlorothiazide (HCTZ) — HCTZ 25mg (Capsule)
Drug: Placebo to Hydrochlorothiazide (HCTZ) — HCTZ 25mg (Capsule) Matching Placebo
Drug: Ramipril — Ramipril 10mg (Tablet)

SUMMARY:
The study is designed to primarily assess the effect of aliskiren on albuminuria in patients with non-diabetic nephropathy when treated with ramipril and volume intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 18 years and above
* Patients with chronic kidney disease of non-diabetic origin
* Glomerular filtration rate >30 ml/min/1.73m2
* Patients with a history of hypertension and msSBP (mean systolic blood pressure) of <160 mm Hg and msDBP (mean diastolic blood pressure) <105 mm Hg at screening and baseline.
* Subjects must have a body mass index (BMI) within the range of 18 and 35 kg/m2

Exclusion Criteria:

* Previously treated (within 3 months of screening) with aliskiren or a combination of aliskiren and ramipril.
* Severe hypertension (msDBP ≥110 mmHg and msSBP ≥180 mmHg)
* Pregnant or nursing (lactating) women,
* A medical history of unstable coronary artery disease, myocardial infarction, coronary bypass surgery or cerebrovascular accident within the last six (6) months
* Diabetes mellitus, Heart failure
* High rate of renal function loss
* History of severe hypersensitivity or contraindications to any of the medications or drugs belonging to the similar therapeutic class as the study drugs and the excipients.
* History of liver disease, positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Netherlands (2):
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leeuwarden

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (Day 1 to End of Week 6)
Arm/Group | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)+HCTZ/Ram+Ali/Ram | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)/Ram+Ali + HCTZ/Ram
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Period 2 (Weeks 7 to 12)
Arm/Group | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)+HCTZ/Ram+Ali/Ram | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)/Ram+Ali + HCTZ/Ram
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Abnormal laboratory value(s) | 0 | 1
Period: Period 3 (Weeks 13 to 18)
Arm/Group | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)+HCTZ/Ram+Ali/Ram | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)/Ram+Ali + HCTZ/Ram
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Period 4 (Weeks 19 to 26)
Arm/Group | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)+HCTZ/Ram+Ali/Ram | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)/Ram+Ali + HCTZ/Ram
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)+HCTZ/Ram+Ali/Ram | Ramipril (Ram) +HCTZ/Ram+Aliskiren (Ali)/Ram+Ali + HCTZ/Ram | Total
Number analyzed (Participants) | 4 | 4 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 50.5 (6.76) | 58.5 (8.70) | 54.5 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Effect of Aliskiren on Albuminuria as Measured by Urinary Albumin Excretion Rate (UAER)
Description: Two 24-hour collections of urine were to be made at each study visit. The arithmetic mean of the two collections were planned to be used in the calculation of summary statistics and the statistical analyses.
Time Frame: 26 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Groups:
- Ramipril +HCTZ: All patients were treated for 6 weeks with daily doses of ramipril 10 mg + placebo to 2 x 150 mg aliskiren (300 mg) + HCTZ 25 mg
- Ramipril+Aliskiren + HCTZ: All patients were treated for 6 weeks with daily doses of ramipril 10 mg + aliskiren 300 mg* (2 x 150 mg) + HCTZ 25 mg
  * Patients were started on aliskiren 150 mg for the 1st week and up-titrated to 300 mg (2 x 150 mg) at the beginning of the 2nd week and continued on this dose until the end of the 6th week of the period
- Ramipril+Aliskiren: All patients were treated for 6 weeks with daily doses of ramipril 10 mg + aliskiren 300 mg* (2 tablets of 150 mg) + placebo to 25 mg HCTZ
  *Patients were started on aliskiren 150 mg for the 1st week and up-titrated to 300 mg (2 x 150 mg) at the beginning of the 2nd week and continued on this dose until the end of the 6th week of the period
- Ramipril: All patients were treated for 8 weeks with daily doses of ramipril 10 mg + placebo to 2 x 150 mg aliskiren + placebo to 25 mg HCTZ
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Effect of Aliskiren on Albuminuria as Measured by Creatinine Indexed Albumin
Description: as for outcome 1
Time Frame: 26 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean Sitting Systolic Blood Pressure (msSBP)
Description: At study entry, blood pressure (BP) was measured in both arms. If there was a clinically relevant difference in readings between arms (≥ 10 mmHg in systolic BP and/or ≥ 5 mmHg in diastolic BP), the arm with higher BP reading was used. If there was no clinically significant difference between arms, the non-dominant arm was used through out study. Systolic blood pressure were assessed after the patient rested quietly in the sitting position for at least 3 minutes. For each sitting assessment, blood pressure was assessed at least 3 times. From these assessments, msSBP was calculated. All BP measurements were to be performed on the same arm.
Time Frame: 26 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Mean Sitting Diastolic Blood Pressure (msDBP)
Description: At study entry, blood pressure (BP) was measured in both arms. If there was a clinically relevant difference in readings between arms (≥ 10 mmHg in systolic BP and/or ≥ 5 mmHg in diastolic BP), the arm with higher BP reading was used. If there was no clinically significant difference between arms, the non-dominant arm was used through out study. Diastolic blood pressure were assessed after the patient rested quietly in the sitting position for at least 3 minutes. For each sitting assessment, blood pressure was assessed at least 3 times. From these assessments, msDBP was calculated. All BP measurements were to be performed on the same arm.
Time Frame: 26 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Mean Glomerular Filtration Rate (GFR) as Measurement of Renal Function
Description: All patients had to visit the main center for renal function measurements. The measurements were performed using the constant infusion method with I-iothalamate (IOT) and I-hippuran. GFR was calculated as the urinary clearance of IOT.
Time Frame: 26 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Mean Effective Renal Plasma Flow (ERPF) as One of Hemodynamic Assessments
Time Frame: 26 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Renal Filtration Fraction (RFF) as One of Hemodynamic Assessments
Time Frame: 26 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Mean Extracellular Volume (ECV) as One of Hemodynamic Assessments
Time Frame: 26 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Plasma Rennin Activity (PRA)
Description: Blood biomarkers were obtained from blood samples in all patients at the time points such as baseline, week 6, week 12, week 18 and week 26. Plasma PRA is a direct measure of the formation of Ang I in the plasma.
Time Frame: Baseline to week 26
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Plasma Rennin Concentration (PRC)
Description: Blood biomarkers were obtained from blood samples in all patients at the time points such as baseline, week 6, week 12, week 18 and week 26. PRC measures the concentration of immunoactive renin in the plasma.
Time Frame: Baseline to week 26
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Death as Assessment of Safety and Tolerability of Aliskiren Added to Ramipril
Time Frame: 26 weeks
Population: The safety analysis set consisted of all patients who received at least one study drug and had no major protocol deviations that could have impacted safety data.
Measure: Number; unit: Participants
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Number analyzed (Participants) | 8 | 7 | 7 | 6
Participants
  patients with adverse events | 7 | 5 | 3 | 4
  patients with serious adverse events | 0 | 0 | 0 | 0
  patients with death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ramipril +HCTZ | Ramipril+Aliskiren + HCTZ | Ramipril+Aliskiren | Ramipril
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 7/8 | 5/7 | 3/7 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ramipril +HCTZ (N=8) | Ramipril+Aliskiren + HCTZ (N=7) | Ramipril+Aliskiren (N=7) | Ramipril (N=6)
Fatigue (General disorders) | 3 | 2 | 2 | 2
Dizziness (Nervous system disorders) | 4 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Edema peripheral (General disorders) | 1 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Renal function test abnormal (Investigations) | 0 | 0 | 1 | 0
Salt craving (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.